CLINICAL TRIAL: NCT06989736
Title: Evaluation of Taste Sensation Changes in Individuals Undergoing Fixed Orthodontic Treatment
Brief Title: Evaluation of Taste Sensation Changes During Fixed Orthodontic Treatment
Acronym: TASTEFIXED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Sinem Kuru Kaygun, PhD student, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-KAEK-79-23-10
Record Dates: First submitted 2025-05-13; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Taste Disorders; Orthodontic Appliance Complication; Malocclusion
MeSH Terms: conditions — Taste Disorders; Malocclusion

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either a fixed orthodontic treatment group or a no-treatment control group in parallel, and taste perception changes were compared between these groups over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): 64 individuals who commenced fixed orthodontic treatment will gargle with the 9 different taste solutions for 15 seconds and then be asked whether they perceive the taste.
  Interventions: Diagnostic Test: Taste Test
- Control group (Other): Participants receiving no orthodontic treatment; monitored for taste perception at the same time intervals.
  Interventions: Diagnostic Test: Taste Test

INTERVENTIONS:
Diagnostic Test: Taste Test — Participants received nine solutions (tasteless, sweet, salty, sour, and bitter; each in two concentrations) before treatment and six weeks later.

SUMMARY:
The aim of this study is to determine the changes in taste perception that may occur before and after the initiation of treatment in patients undergoing fixed orthodontic treatment. A total of 128 patients from Biruni University Faculty of Dentistry, Orthodontics Clinic, were randomly selected to either a fixed orthodontic treatment group (n=64) or a control group (n=64), Taste sensation was assessed using nine solutions representing different taste modalities (sweet, salty, sour and bitter), with evaluations conducted via a Visual Analog Scale (VAS) before treatment and six weeks post-treatment. Statistical analyses were performed using the Mann-Whitney U test, Wilcoxon Signed-Rank test and Pearson Chi-Square test. The study found statistically significant differences in sweet taste perception between the first and second sessions in the low-dose experimental group and in bitter taste perception in the high-dose experimental group (p<0.05). However, no statistically significant differences were observed between the experimental and control groups across all taste types and time points (p>0.05). While orthodontic treatment resulted in some changes in sweet and bitter taste perception, no overall significant differences were found between the experimental and control groups. Increased salivary flow rate during treatment and good oral hygiene may help minimize potential effects on taste perception.

DETAILED DESCRIPTION:
This interventional clinical study aimed to investigate whether fixed orthodontic treatment affects taste perception in adolescent patients. A total of 128 participants aged 10 to 19 years were recruited and randomly assigned to either a fixed orthodontic treatment group or a control group. Exclusion criteria included systemic diseases, smoking, medications affecting taste, and salivary gland disorders.

Taste perception was assessed using nine standard solutions representing sweet, salty, sour, and bitter tastes at two concentrations each, plus a tasteless solution (distilled water). Evaluations were performed using a Visual Analog Scale (VAS) before treatment and six weeks after treatment initiation.

The study received ethical approval from the Biruni University Interventional Clinical Research Ethics Committee (Decision No: 2015-KAEK-79-23-10). Informed consent was obtained from all participants or their guardians.

Statistical analyses revealed significant intra-group differences in sweet and bitter taste perceptions in the experimental group, while no significant inter-group differences were found across time points. These findings suggest that fixed orthodontic treatment may cause temporary changes in certain taste perceptions, which could be mitigated by increased salivary flow and good oral hygiene practices.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 19 years
* Applied to the Orthodontics Clinic at Biruni University Faculty of Dentistry
* Provided written informed consent (or assent with guardian consent if under 18)
* Randomized to either fixed orthodontic treatment or control group

Exclusion Criteria:

* Presence of systemic disease
* Current smoker
* Using medications known to affect taste (e.g., captopril, fluoxetine hydrochloride, sulfadoxine)
* Diagnosed with salivary gland disorders
* Presence of any pathology that may cause dry mouth (xerostomia)

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Taste Perception Score | From baseline (pre-treatment) to 6 weeks post-treatment
  Taste perception was measured using a Visual Analog Scale (VAS) across four taste modalities (sweet, salty, sour, bitter). VAS scores (0-100) were compared between baseline and 6 weeks post-treatment.

SECONDARY OUTCOMES:
Comparison of Taste Perception Between Treatment and Control Groups | 6 weeks post-treatment
  Evaluation of differences in taste perception scores (VAS) across treatment and control groups after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Asli Konca Taşova, DDS, PhD, Study Chair — Uskudar University Faculty of Dentistry, Department of Orthodontics
Locations (1):
- Biruni University Faculty of Dentistry Department of orthodontic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study protocol and ethics committee approval do not include provisions for data sharing

REFERENCES:
- [Derived] Kuru Kaygun S, Konca Tasova FA. Effects of fixed orthodontic treatment on taste perception: a randomized controlled trial. Clin Oral Investig. 2025 Dec 19;30(1):17. doi: 10.1007/s00784-025-06714-6. PMID 41417250